CLINICAL TRIAL: NCT03757715
Title: The Role of Regional Anesthesia to Reduce Opioid Requirements Following Functional Endoscopic Sinus Surgery (FESS)
Brief Title: Regional Anesthesia to Reduce Opioid Use Following Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Brad Woodworth, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-300000567
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): 20 mL of 1.3% bupivacaine with 2 mg dexamethasone injected locally in the location for sensory nerves of the sinus cavities and face during the functional endoscopic sinus surgery (FESS) procedure
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone
- Control Group (No Intervention): No regional anesthetic of any kind during the functional endoscopic sinus surgery (FESS) procedure

INTERVENTIONS:
Drug: Bupivacaine — 20 mL of 1.3% bupivacaine
  Other Names: Marcaine
  Arms: Treatment Group
Drug: Dexamethasone — 2 mg dexamethasone
  Other Names: Ozurdex
  Arms: Treatment Group

SUMMARY:
Opioids are prescribed for moderate to severe pain disorders; however, there are contraindications and side effects that are common to all opioids. The investigators hypothesize using regional anesthetic during sinus surgery will reduce surgical pain, therefore decreasing the need for post-operative opioid medication. The primary of objective is to determine if a long-acting local regional anesthetic applied during a surgery will reduce post-operative oral opioid usage.

DETAILED DESCRIPTION:
Opioid analgesics are prescribed for moderate to severe acute pain; however, there are contraindications, cautions, and side effects that are common with all opioids. Dependence and tolerance are also likely with regular opioid use, resulting in the current nationwide opioid epidemic. In Alabama alone, there were 343 opioid-related overdose deaths in 2016, 124 of which were related to prescription opioids. Alabama providers have the highest prescribing rate in the country, nearly twice the national rate, per the NIH/NIDA website. In 2015, the Centers for Disease Control (CDC) released prescribing guidelines relating to chronic pain, and in 2018 Alabama's Blue Cross/Blue Shield insurance group limited the supply of opioids allowed to their members to 7 days.

There is currently no clinical guideline for prescribing post operative opioid medications for functional endoscopic sinus surgery (FESS). A 2018 survey documenting prescribing patterns by 168 members of the American Rhinologic Society found that most physicians who participated prescribed, on average, 27 opioid pain pills for patients after surgery. Prior studies have been performed to help decrease the pain patient's feel after sinus surgery. Haytoglu in 2016 revealed that adding non-absorbable sinus packs loaded with local anesthetics such as bupivacaine achieved less pain values and improved patient satisfaction scores.

Given this current data the investigators believe injecting patients with a long acting analgesic during the procedure will help reduce post-operative pain. If the investigators can decrease the amount of pain patients have in the post-operative period, they can theoretically decrease the number of opioid pain pills prescribed. The investigators plan to also track the number of opioid pills consumed by patients in the post-operative period to obtain a somewhat uniform prescribing pattern within surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to sign informed consent form
* Able to comply with all study procedures and availability for the duration of the study
* Able to speak English
* Diagnosis of chronic rhinosinusitis
* Scheduled to receive functional endoscopic sinus surgery (FESS) at UAB

Exclusion Criteria:

* Current use of opioid medication
* Known allergic reactions to components of the study intervention
* History of IV drug use or abuse
* History of opioid abuse
* History of chronic pain disorder
* Treatment with another investigational drug or other intervention within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Woodworth, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were excluded prior to assignment.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 21 | 25
Completed | 16 | 15
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 4 | 9
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.69 (17.79) | 36.73 (13.10) | 42.90 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.19 (7.66) | 31.71 (11.10) | 31.44 (9.32)
Diabetes [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 4
  No | 15 | 12 | 27
Anxiety/Depression [Count of Participants; unit: Participants]
  No | 11 | 14 | 25
  Yes | 5 | 1 | 6
Migraine [Count of Participants; unit: Participants]
  No | 15 | 12 | 27
  Yes | 1 | 3 | 4
Obstructive Sleep Apnea [Count of Participants; unit: Participants]
  No | 14 | 12 | 26
  Yes | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Participant Pain Control
Description: Self-report of pain score on a scale of 0 to 10, with 0 being "no pain" and 10 being "worst pain imaginable"
Time Frame: 10 days
Population: Both groups were analyzed on the average number of pain pills taken during the post-operative time and average pain scores per day postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 16 | 15
units on a scale
  POD 0 | 4.5 (2.83) | 5.87 (2.85)
  POD1 | 4.63 (1.86) | 5.00 (1.96)
  POD 2 | 4.06 (1.84) | 4.13 (1.89)
  POD 3 | 4.13 (1.46) | 3.20 (2.01)
  POD 4 | 3.38 (1.93) | 2.67 (2.02)
  POD 5 | 3.00 (2.42) | 2.33 (1.76)
  POD 6 | 3.00 (2.58) | 2.2 (1.7)
  POD 7 | 2.56 (2.45) | 2.13 (1.6)
  POD 8 | 2.13 (2.45) | 1.67 (1.76)
  POD 9 | 2.19 (2.34) | 1.73 (2.22)
  POD 10 | 2.13 (2.50) | 1.27 (2.21)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.16, t-test, 1 sided

2. Secondary Outcome: Opioid Medication Use
Description: Amount of opioid medication used, based on pill count
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: pills consumed
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 16 | 15
pills consumed
  POD 0 | 1.38 (1.03) | 1.07 (1.22)
  POD 1 | 2.31 (1.40) | 1.87 (1.92)
  POD 2 | 1.69 (1.66) | 1.40 (1.81)
  POD 3 | 1.63 (1.45) | 1.07 (1.39)
  POD 4 | 0.97 (1.49) | 1.00 (1.36)
  POD 5 | 0.594 (1.11) | 0.567 (1.23)
  POD 6 | 0.50 (1.09) | 0.30 (0.79)
  POD 7 | 0.38 (0.885) | 0.27 (0.799)
  POD 8 | 0.25 (0.577) | 0.20 (0.775)
  POD 9 | 0.31 (0.60) | 0.27 (1.03)
  POD 10 | 0.31 (0.60) | 0.27 (0.80)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.42, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT03757715/Prot_ICF_004.pdf